CLINICAL TRIAL: NCT04812210
Title: Quality of Life and Neurodevelopment Assessment of Children With Congenital Heart Disease Aged 2 to 4 Years : a Multicentre Controlled Cross-sectional Study
Brief Title: Quality of Life and Neurodevelopment Assessment of Children With Congenital Heart Disease Aged 2 to 4 Years
Acronym: QoLCHD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University of Montpellier - Inserm 1046 - PhyMeddExp (Unknown); Saint Pierre Institute - Palavas les Flots (Unknown); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0083
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Congenital Heart Disease
Keywords: health related quality of life; pediatrics; cardiology
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: children with congenital heart disease aged 2 to 4 years.: case: children with congenital heart disease aged 2 to 4 years.
- control children recruited in kindergartens and schools aged 2 to 4 years: control children recruited in kindergartens and schools aged 2 to 4 years

SUMMARY:
Congenital heart diseases (CHD) are the firt cause of congenital malformations (8 for 1000 births). Since the 90's, great advances in prenatal diagnosis, pediatric cardiac surgery, intensive care, and cardiac catheterization have reduced morbidity and early mortality in this population. Nowadays, health-related quality of life (HRQoL) assessment of this population is in the foreground. Our team is a tertiary care center for management of patients with CHD, from the fetal period to adulthood. The investigators have been conducting a clinical research program on HRQoL in pediatric and CHD. The investigators thus demonstrated the link between cardiopulmonary fitness and HRQoL in children with CHD aged 8 to 18 years, the correlation between functional class and HRQoL in adults with CHD, the impact of therapeutic education on HRQoL in children under anticoagulants and the lack of difference between the HRQoL of children CHD aged 5 to 7 years old and that of control children. Currently, no controlled cross-sectional quality of life study assessment has been leded in the youngest children with CHD. This present study therefore extends our work in younger children aged 2 to 4 years.

DETAILED DESCRIPTION:
248 patients will be enrolled in this study (124 children in each group).

Patients from group 1 will be included during their annual medical check-up. HRQoL questionnaire, neurodevelopmental status scale and clinical status will be assessed during this site visit. No supplementary visit, directly related to the research, will be necessary. Three sites will participate to the study, members of he French national network for complex congenital heart diseases (M3C) .

Participants (healthy children) from group 2 will be included from kindergartens and schools. The prior agreement of the Ministry of National Education will be obtained before any procedure related to this study.

ELIGIBILITY:
Inclusion criteria:

* Children aged 2 to 4 years old.
* Group 2 : Chldren with CHD (as defined in the ACC-CHD classification).

Exclusion criteria:

* Other comorbidity affecting quality of life (polymalformative syndrome, extracardiac organ failure, severe genetic disease).
* Surgical procedure during the last 6 months.
* Inability to understand the HRQoL questionnaire (parents) :non-french speaker, severe intellectual disability.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Groupe 1 : Children with congenital heart disease aged 2 to 4 years Groupe 2 : Healthy children aged 2 to 4 years
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the total score of the proxy HRQoL questionnaire | 1 day
  Comparison of the total score of the proxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) between patients with CHD and control children : The proxy HRQoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 demensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed.

SECONDARY OUTCOMES:
Comparison of score by dimensions of the proxy HRQoL questionnaire | 1 day
  Comparison of score by dimensions of the proxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) between patients with CHD and schoolchildren aged 2 to 4 years : The proxy HRQoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 demensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order o get score by dimensions of scale we must sum the items scores over the number of items answered. If more than 50% of the items in the scale are missing, the scale scores should not be computed.
Comparison of score of the roxy HRQoL questionnaire | 1 day
  Comparison of score of the roxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the type of the CHD unsing the ACC-CHD classification : The proxy HRQoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed.
Comparison of score of the proxy HRQoL questionnaire | 1 day
  Comparison of score of the proxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the severity of the CHD unsing the BETHESDA classification : The proxy HRQoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 demensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be
Comparison of score of the HRQoL questionnaire | 1 day
  Comparison of score of the HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the patient functional status unsing the Ross classification : The proxy HRQoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 demensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be
Comparison of score of the proxy HRQoL questionnaire | 1 day
  Comparison of score of the proxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the prognostic classification of the CHD unsing Davey B.T classification : The proxy HRQoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 demensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be
Study of the association of the following variables related to the patient and to the CHD with the scores of the proxy HRQoL questionnaire | 1 day
  Study of the association of the following variables related to the patient and to the CHD with the scores of the proxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) . Univariate end multivariate analysis will be performed. The variables are:
  * sex of the patient,
  * age at diagnosis of CHD (pre or post natal)
  * cardiac clinical data
  * neurodevelopmental status
Evaluation of the psychometric properties of the proxy HRQoL questionnaire | 1 day
  Evaluation of the psychometric properties of the proxy HRQoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) . for children aged 2 to 4 years old : The Pediatric Quality of Life Inventory Version 4.0 (PedsQLTM 4.0) is a questionnaire widely used in pediatric clinical trials. This questionnaire was translated and linguistically validated in French, but no complete psychometric validation for French children aged 2 to 4 years has been performed yet. Reliability and validity are considered the main measurement properties of such instruments

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER; Johanna Calderon, Study Chair — PhyMeddExp; Sophie Guillaumont, Principal Investigator — Saint Pierre Institute - Palavas les Flots; Jean-Benoit Thmabo, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC